CLINICAL TRIAL: NCT01778556
Title: Short Term Effects of Leptin Withdrawal or Initiation in Lipodystrophy Independent of Energy Intake
Brief Title: Short-term Effects of Leptin in People With Lipodystrophy
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: 130057; 13-DK-0057
Record Dates: First submitted 2013-01-26; First posted 2013-01-29 (Estimated); Results first posted 2019-11-13 (Actual); Last update posted 2019-11-13 (Actual); Status verified 2019-02-25

CONDITIONS: Lipodystrophy
Keywords: Lipodystrophy; Leptin; Energy Expenditure; Diabetes; Hypertriglyceridemia
MeSH Terms: conditions — Lipodystrophy; Diabetes Mellitus; Hypertriglyceridemia | interventions — metreleptin

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes

ARMS (2):
- Leptin naive (Experimental): Studied for 5 days without metreleptin, then 14 days while taking metreleptin
  Interventions: Biological: Metreleptin
- On-leptin (Experimental): Studied for 5 days while taking metreleptin, then 14 days during metreleptin withdrawal
  Interventions: Biological: Metreleptin

INTERVENTIONS:
Biological: Metreleptin — Recombinant analog of the human hormone, leptin

SUMMARY:
Background:

- Lipodystrophy is a condition where people do not have enough fat in the body. People with lipodystrophy can have problems such as diabetes or an enlarged liver. Researchers are looking at how leptin, a hormone produced by fat cells, can help people with these problems. Leptin helps control appetite and how the body stores food. Taking leptin can help people with lipodystrophy eat less food, which may help treat diabetes and other problems. To better understand how leptin works, researchers want to do an inpatient study on leptin treatment in people with lipodystrophy.

Objectives:

- To study how leptin treatment affects lipodystrophy.

Eligibility:

- Individuals between 14 and 70 years of age who have lipodystrophy.

Design:

* All participants will have a 19-day stay at the National Institutes of Health Clinical Center. One group of participants will have tests for 5 days before starting to take leptin. They will then take leptin for 2 weeks, and have more tests. The other group of participants will have tests for 5 days while taking leptin. They will then take stop taking leptin for 2 weeks, and have more tests, and then they will start taking leptin again.
* Participants will have regular blood and urine tests during the visit. Some of the blood tests will look at insulin levels. Some will look at how the body metabolizes sugar and fat. Other tests will check hormone levels, especially of reproductive hormones.
* During the visit, participants will spend 3 separate days in a metabolic chamber, a special room that measures how many calories the body uses. Urine samples will be collected during these stays.
* Participants will also have several body imaging studies, including magnetic resonance imaging and a body composition scan.
* Physical activity will be tested with an exercise bicycle and an electronic activity monitor.
* Participants will be asked questions about hunger and comfort levels throughout the stay.

DETAILED DESCRIPTION:
Background

Leptin is an adipocyte-derived hormone that can be thought of as a signal from adipose tissue to the rest of the body conveying information about long-term nutritional status. Patients with lipodystrophy have leptin deficiency secondary to lack of adipose tissue, and thus represent a natural model for studying the effects of leptin deficiency and replacement in humans. Leptin replacement in lipodystrophy ameliorates metabolic and endocrine abnormalities, including reducing food intake, improving insulin resistance and diabetes, reducing ectopic lipid, and normalizing reproduction. The reduction in energy intake induced by leptin replacement is likely responsible for part of the improvements observed in glucose and lipid metabolism. The clinical effects of leptin that are independent of changes in energy intake, and the mechanisms underlying these effects, have been poorly explored in humans.

Aim

The primary aim of this study is to determine the energy intake-independent effects of leptin on energy metabolism in lipodystrophic subjects. The major aspects of energy metabolism to be studied are:

1. Lipid metabolism, including fasting lipids, lipolysis and fatty acid turnover, and ectopic lipid storage.
2. Glucose metabolism, including fasting glucose, endogenous glucose production, and insulin sensitivity
3. Energy expenditure, including total and resting energy expenditure, skeletal muscle work efficiency, and spontaneous physical activity

In addition, the effects of leptin on endocrine and autonomic function will be examined, including effects on the thyroid, gonadal, and adrenal axes, as well as blood pressure, body temperature, and heart rate variability.

Methods

This is a non-randomized, parallel group study. Two groups of patients aged 14 to 70 years with lipodystrophy will be studied: leptin naive and leptin treated. Minors will only be included in the leptin naive arm. All subjects will be stabilized on a weight maintenance diet for 5 days (Period 1). After this, leptin will be withdrawn from leptin treated subjects, and leptin will be initiated in leptin naive subjects for a period of 14 days (Period 2). The same isocaloric diet will be continued throughout both Periods, permitting study of leptin s effects independent of energy intake.

All subjects will undergo metabolic testing on admission, at the end of Period 1, and throughout Period 2, to generate a detailed short-term time course of the effects of leptin initiation or withdrawal. At the end of Period 2, leptin will be continued in the leptin naive subjects, and restarted in the leptin treated subjects. Repeat metabolic testing will be performed 6-12 months after leptin initiation in the leptin-naive cohort to generate information on leptin s long-term effects.

ELIGIBILITY:
* INCLUSION CRITERIA:
* Age 14-70 years (children under age 18 will only be enrolled in the leptin-naive arm of the study
* Clinically-significant lipodystrophy as defined in protocol 02-DK-0022 (Long Term Efficacy of Leptin Replacement in the Treatment of Lipodystrophy). Relevant inclusion criteria for enrollment in protocol 02-DK-0022 are (summarized):

  * Lipodystrophy identified by the study physician during physical examination as an absence of fat outside the range of normal
  * Circulating leptin levels < 12.0 ng/mL in females and < 8.0 ng/mL in males
  * Presence of at least one of the following metabolic abnormalities:

    1. Diabetes as defined by the 2007 American Diabetes Association criteria
    2. Fasting insulin >30 microU/mL
    3. Fasting hypertriglyceridemia >200 mg/dL
* Co-enrolled in protocol 02-DK-0022 and either:

  * Leptin naive, with plans to initiate leptin treatment during the current study. For the purpose of this study, leptin naive will be defined as having received no exogenous leptin in the 4 months prior to study participation. Thus, subjects who previously received leptin therapy, discontinued, and wish to restart are eligible.

Or

--Leptin treated, meaning the subject has taken a stable dose of exogenous leptin for a minimum of 4 months (adults over age 18, only)

EXCLUSION CRITERIA:

In leptin treated subjects only, the following exclusion criteria apply:

* Poorly controlled diabetes at study entry (hemoglobin A1c greater than or equal to 9%)
* Poorly controlled hypertriglyceridemia at study entry (serum triglycerides > 800 mg/dL)
* Extreme hypertriglyceridemia prior to leptin (triglycerides greater than 2000 mg/dL at initiation of leptin treatment)
* History of chronic or recurrent acute pancreatitis (> 1 episode), or a single episode of pancreatitis while receiving leptin treatment
* Lipase greater than the upper limit of normal (491 units/L) at study entry

In all subjects (leptin treated and leptin naive), the following exclusion criteria apply:

* Known HIV infection or HIV-associated lipodystrophy
* History of diabetic ketoacidosis
* Active inflammatory disease (e.g. dermatomyositis)
* Change in diabetes or lipid-lowering medications within the past 6 weeks
* Estimated glomerular filtration rate < 30 mL/minute
* Current or recent (past 2 weeks) use of systemic glucocorticoids
* Inadequately controlled hypothyroidism (TSH < 0.4 or >4 mcIU/L) or change in thyroid medication in the past 8 weeks.
* Pregnancy or breast-feeding
* Psychiatric disorder impeding competence or compliance
* Any medical condition or medication that will increase risk to the subject (e.g. ischemic heart disease, decompensated liver disease) or that will interfere with interpretation of study data (e.g. Cushing s syndrome).

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2013-01-26; Primary Completion 2018-02-23 (Actual); Study Completion 2018-02-23 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Rebecca J Brown, M.D., Principal Investigator — National Institute of Diabetes and Digestive and Kidney Diseases (NIDDK)
Locations (1):
- National Institutes of Health Clinical Center, 9000 Rockville Pike, Bethesda, Maryland, United States

REFERENCES:
- [Background] Ahima RS, Dushay J, Flier SN, Prabakaran D, Flier JS. Leptin accelerates the onset of puberty in normal female mice. J Clin Invest. 1997 Feb 1;99(3):391-5. doi: 10.1172/JCI119172. PMID 9022071
- [Background] Ahima RS, Prabakaran D, Mantzoros C, Qu D, Lowell B, Maratos-Flier E, Flier JS. Role of leptin in the neuroendocrine response to fasting. Nature. 1996 Jul 18;382(6588):250-2. doi: 10.1038/382250a0. PMID 8717038
- [Background] Chehab FF, Lim ME, Lu R. Correction of the sterility defect in homozygous obese female mice by treatment with the human recombinant leptin. Nat Genet. 1996 Mar;12(3):318-20. doi: 10.1038/ng0396-318. PMID 8589726
- [Derived] Quaye E, Chacko S, Startzell M, Brown RJ. Leptin Decreases Gluconeogenesis and Gluconeogenic Substrate Availability in Patients With Lipodystrophy. J Clin Endocrinol Metab. 2023 Dec 21;109(1):e209-e215. doi: 10.1210/clinem/dgad445. PMID 37515588
- [Derived] Meral R, Malandrino N, Walter M, Neidert AH, Muniyappa R, Oral EA, Brown RJ. Endogenous Leptin Concentrations Poorly Predict Metreleptin Response in Patients With Partial Lipodystrophy. J Clin Endocrinol Metab. 2022 Mar 24;107(4):e1739-e1751. doi: 10.1210/clinem/dgab760. PMID 34677608
- [Derived] Nguyen ML, Sachdev V, Burklow TR, Li W, Startzell M, Auh S, Brown RJ. Leptin Attenuates Cardiac Hypertrophy in Patients With Generalized Lipodystrophy. J Clin Endocrinol Metab. 2021 Oct 21;106(11):e4327-e4339. doi: 10.1210/clinem/dgab499. PMID 34223895
- [Derived] Grover A, Quaye E, Brychta RJ, Christensen J, Startzell MS, Meehan CA, Valencia A, Marshall B, Chen KY, Brown RJ. Leptin Decreases Energy Expenditure Despite Increased Thyroid Hormone in Patients With Lipodystrophy. J Clin Endocrinol Metab. 2021 Sep 27;106(10):e4163-e4178. doi: 10.1210/clinem/dgab269. PMID 33890058
- [Derived] Baykal AP, Parks EJ, Shamburek R, Syed-Abdul MM, Chacko S, Cochran E, Startzell M, Gharib AM, Ouwerkerk R, Abd-Elmoniem KZ, Walter PJ, Walter M, Muniyappa R, Chung ST, Brown RJ. Leptin decreases de novo lipogenesis in patients with lipodystrophy. JCI Insight. 2020 Jul 23;5(14):e137180. doi: 10.1172/jci.insight.137180. PMID 32573497
- [Derived] Sekizkardes H, Chung ST, Chacko S, Haymond MW, Startzell M, Walter M, Walter PJ, Lightbourne M, Brown RJ. Free fatty acid processing diverges in human pathologic insulin resistance conditions. J Clin Invest. 2020 Jul 1;130(7):3592-3602. doi: 10.1172/JCI135431. PMID 32191645
- [Derived] Sekizkardes H, Cochran E, Malandrino N, Garg A, Brown RJ. Efficacy of Metreleptin Treatment in Familial Partial Lipodystrophy Due to PPARG vs LMNA Pathogenic Variants. J Clin Endocrinol Metab. 2019 Aug 1;104(8):3068-3076. doi: 10.1210/jc.2018-02787. PMID 31194872
- [Derived] Brown RJ, Valencia A, Startzell M, Cochran E, Walter PJ, Garraffo HM, Cai H, Gharib AM, Ouwerkerk R, Courville AB, Bernstein S, Brychta RJ, Chen KY, Walter M, Auh S, Gorden P. Metreleptin-mediated improvements in insulin sensitivity are independent of food intake in humans with lipodystrophy. J Clin Invest. 2018 Aug 1;128(8):3504-3516. doi: 10.1172/JCI95476. Epub 2018 Jul 16. PMID 29723161
- [Derived] Brown RJ, Meehan CA, Cochran E, Rother KI, Kleiner DE, Walter M, Gorden P. Effects of Metreleptin in Pediatric Patients With Lipodystrophy. J Clin Endocrinol Metab. 2017 May 1;102(5):1511-1519. doi: 10.1210/jc.2016-3628. PMID 28324110
- See also: NIH Clinical Center Detailed Web Page — https://clinicalstudies.info.nih.gov/cgi/detail.cgi?B_2013-DK-0057.html

RESULTS

PARTICIPANT FLOW:
Period: Intervention 1 (5 Days)
Arm/Group | Leptin Naive | On-leptin
Started | 15 | 10
Completed | 15 | 8
Not Completed | 0 | 2
Not completed — Protocol Violation | 0 | 1
Not completed — Withdrawal by Subject | 0 | 1
Period: Intervention 2 (14 Days)
Arm/Group | Leptin Naive | On-leptin
Started | 15 | 8
Completed | 14 | 8
Not Completed | 1 | 0
Not completed — Protocol Violation | 1 | 0
Period: Long-term Follow-up
Arm/Group | Leptin Naive | On-leptin
Started | 15 | 0 (no long-term follow-up period in on-leptin arm)
Completed | 14 | 0 (no long-term follow-up period in on-leptin arm)
Not Completed | 1 | 0
Not completed — noncompliance with metreleptin | 1 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Leptin Naive | On-leptin | Total
Number analyzed (Participants) | 15 | 8 | 23
Age, Continuous [Mean (Standard Deviation); unit: years] | 32 (17) | 25 (6) | 28 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 5 | 17
  Male | 3 | 3 | 6
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  White | 9 | 4 | 13
  Hispanic | 4 | 2 | 6
  African American | 0 | 2 | 2
  Asian | 1 | 0 | 1
  Other | 1 | 0 | 1
Type of lipodystrophy [Count of Participants; unit: Participants]
  Generalized | 3 | 8 | 11
  Partial | 12 | 0 | 12
Subtype of lipodystrophy [Count of Participants; unit: Participants]
  Congenital generalized lipodystrophy | 3 | 7 | 10
  Familial partial lipodystrophy | 12 | 0 | 12
  Acquired generalized lipodystrophy | 0 | 1 | 1
Endogenous leptin level [Mean (Standard Deviation); unit: ng/dl] | 9.5 (10.2) | 1.2 (0.5) | 7.4 (10.1)

OUTCOME MEASURES:

1. Primary Outcome: Total Body Insulin Sensitivity
Description: Total body insulin sensitivity (measured as glucose disposal rate during a hyperinsulinemic, euglycemic clamp)
Time Frame: Intervention 1 (5 days), Intervention 2 (14 days), and Long-term follow-up (6 months)
Population: One patient at Period 2 (14 days) in Leptin naive arm was withdrew due to protocol violation.
Measure: Mean (Standard Deviation); unit: mg/kg fat-free mass/min
Arm/Group | Leptin Naive | On-leptin
Number analyzed (Participants) | 15 | 8
mg/kg fat-free mass/min
  Intervention 1 (5 days) | 4.4 (2.3) | 10.9 (4.1)
  Intervention 2 (14 days): number analyzed (Participants) | 14 | 8
  Intervention 2 (14 days) | 5.8 (2.2) | 6.4 (1.8)
  Long-term follow-up (6 months): number analyzed (Participants) | 13 | 0
  Long-term follow-up (6 months) | 8.0 (4.0) |

2. Secondary Outcome: Insulin-mediated Suppression of Hepatic Glucose Production
Description: Hepatic insulin sensitivity (measured as suppression of endogenous glucose production during a hyperinsulinemic, euglycemic clamp)
Time Frame: Intervention 1 (5 days), Intervention 2 (14 days), and Long-term follow-up (6 months)
Population: Measurements were not available.
Measure: Mean (Standard Deviation); unit: percentage
Arm/Group | Leptin Naive | On-leptin
Number analyzed (Participants) | 14 | 8
percentage
  Intervention 1 (5 days): number analyzed (Participants) | 12 | 6
  Intervention 1 (5 days) | 61.2 (23.4) | 77.1 (42.7)
  Intervention 2 (14 days): number analyzed (Participants) | 12 | 6
  Intervention 2 (14 days) | 75.2 (33.1) | 63.8 (31.7)
  Long-term follow-up (6 months): number analyzed (Participants) | 14 | 0
  Long-term follow-up (6 months) | 85.6 (17.9) |

3. Secondary Outcome: Endogenous Rate of Appearance of Palmitate
Description: Endogenous Rate of Appearance of Palmitate is measured in plasma.
Time Frame: Intervention 1 (5 days), Intervention 2 (14 days), and Long-term follow-up (6 months)
Population: Measurements were not available.
Measure: Mean (Standard Deviation); unit: μmol/kg fat-free mass/min
Arm/Group | Leptin Naive | On-leptin
Number analyzed (Participants) | 14 | 8
μmol/kg fat-free mass/min
  Intervention 1 (5 days): number analyzed (Participants) | 11 | 6
  Intervention 1 (5 days) | 3.2 (1.3) | 1.4 (0.7)
  Intervention 2 (14 days): number analyzed (Participants) | 11 | 6
  Intervention 2 (14 days) | 2.8 (1.0) | 1.7 (0.6)
  Long-term follow-up (6 months): number analyzed (Participants) | 14 | 0
  Long-term follow-up (6 months) | 2.2 (0.7) |

ADVERSE EVENTS:
Time Frame: 6 months
Groups:
- Intervention 1 (5 Days) : Leptin Naive: Studied for 5 days without taking metreleptin.
  Metreleptin: Recombinant analog of the human hormone, leptin
- Intervention 2 (14 Days): Leptin Naive: Studied for 14 days while taking metreleptin after the intervention 1 (5 days) : Leptin Naive Metreleptin: Recombinant analog of the human hormone, leptin
- Long-term Follow-up (6 Months): Leptin Naive: Studied for 6 months while taking metreleptin after intervention 2 (14 days): Leptin Naive
  Metreleptin: Recombinant analog of the human hormone, leptin
- Intervention 1 ( 5 Days) : On-Leptin: Studied for 5 days while taking metreleptin
  Metreleptin: Recombinant analog of the human hormone, leptin
- Intervention 1 ( 14 Days): On-Leptin: Studied for 14 days during metreleptin withdrawal after Intervention 1 ( 5 days) : On-Leptin
  Metreleptin: Recombinant analog of the human hormone, leptin
Arm/Group | Intervention 1 (5 Days) : Leptin Naive | Intervention 2 (14 Days): Leptin Naive | Long-term Follow-up (6 Months): Leptin Naive | Intervention 1 ( 5 Days) : On-Leptin | Intervention 1 ( 14 Days): On-Leptin
All-Cause Mortality (participants affected / at risk) | 0/15 | 0/15 | 0/15 | 0/8 | 0/8
Serious Adverse Events (participants affected / at risk) | 0/15 | 1/15 | 2/15 | 0/8 | 0/8
Other Adverse Events (participants affected / at risk) | 0/15 | 2/15 | 4/15 | 0/8 | 0/8
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention 1 (5 Days) : Leptin Naive (N=15) | Intervention 2 (14 Days): Leptin Naive (N=15) | Long-term Follow-up (6 Months): Leptin Naive (N=15) | Intervention 1 ( 5 Days) : On-Leptin (N=8) | Intervention 1 ( 14 Days): On-Leptin (N=8)
abdominal pain of unknown etiology (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA — This adverse event was happened within 30 days window after the end of long-term follow-up.
angioedema secondary to angiotensin- converting enzyme inhibitor use (Cardiac disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA
anemia secondary to menorrhagia (Endocrine disorders) | 0 (0) | 1 (4) | 0 (0) | NA | NA
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Intervention 1 (5 Days) : Leptin Naive (N=15) | Intervention 2 (14 Days): Leptin Naive (N=15) | Long-term Follow-up (6 Months): Leptin Naive (N=15) | Intervention 1 ( 5 Days) : On-Leptin (N=8) | Intervention 1 ( 14 Days): On-Leptin (N=8)
decreased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA
weight loss (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA
hair loss (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA
hypoglycemia (in a subject treated with insulin) (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | NA | NA
injection site reaction (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | NA | NA
menorrhagia (Endocrine disorders) | 0 (0) | 1 (1) | 0 (0) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-14): https://cdn.clinicaltrials.gov/large-docs/56/NCT01778556/Prot_SAP_000.pdf